CLINICAL TRIAL: NCT01813331
Title: ALERT-HF:Adherence to Guidelines in the Treatment of Patients With Chronic Heart Failure
Brief Title: ALERT-HF: Adherence to Guidelines in the Treatment of Patients With Chronic Heart Failure
Acronym: ALERT-HF
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Oliviero Ugo, MD, Federico II University
Other Study IDs: 161/12
Record Dates: First submitted 2013-03-07; First posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

GROUPS / COHORTS (1):
- Chronic Heart Failure Patients: Chronic Heart Failure patients older than 65 years, which accept to participate to the study and give their informed written consent and consecutively refer to the A.R.C.A Campania Cardiologists in the pertaining healthcare districts.

SUMMARY:
ALERT-HF is an observational study aimed to evaluate the diagnostic criteria adopted and the adherence to the current therapeutic guidelines in a large series of patients affected with chronic heart failure. Secondary objective is to evaluate the prevalence of chronic heart failure among all the patients referring to the ambulatory cardiologists of the healthcare district.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heart Failure
* Signature of informed consent
* Age older than 65 years

Exclusion Criteria:

* indication for cardiac surgery or cardiac surgery by less than 3 months
* age less than 65 years
* inability to perform periodic checks
* presence of malignant neoplasms and other severe diseases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Chronic Heart Failure patients older than 65 years, consecutively referred to the A.R.C.A Campania Cardiologists in the pertaining healthcare districts
Sampling Method: Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of patients treated with each of the following indicators of adherence to the current therapeutic guidelines:-ACEI -ARB -beta blockers -loop diuretics -aldosterone antagonists -digoxin -anticoagulant therapy - implantation of cardiac devices | first physical examination and clinical evaluation performed during a 3 months period, from November 2012 to January 2013

SECONDARY OUTCOMES:
evaluate the prevalence of chronic heart failure among all the patients referring to the ambulatory cardiologists of the healthcare district | first evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- ARCA Campania healthcare ambulatories, Naples, Italy